CLINICAL TRIAL: NCT01044355
Title: Effect of Fixed Versus Auto-titrating Continuous Positive Airway Pressure on Blood Pressure and Arterial Stiffness in Patients With Resistant Hypertension and Obstructive Sleep Apnea
Brief Title: Effect of Continuous Positive Airway Pressure (CPAP) Versus Auto-titrating Continuous Positive Airway Pressure (APAP) on Resistant Hypertension (HTN) and Arterial Stiffness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: OSR Medical Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Stella Daskalopoulou, MD, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-038-SDR (SARHT 1001)
Record Dates: First submitted 2010-01-06; First posted 2010-01-07 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Resistant Hypertension; Obstructive Sleep Apnea
Keywords: Resistant Hypertension; Obstructive Sleep Apnea; 24 Hour Blood Pressure; Arterial Stiffness; Insulin Resistance; CPAP; APAP
MeSH Terms: conditions — Sleep Apnea, Obstructive; Insulin Resistance | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- auto-titrating (Active Comparator): Patients being treated for 6 weeks with auto-titrating continuous airway pressure.
  Interventions: Device: APAP
- Fixed (Active Comparator): Patients receiving 6 weeks of treatment with fixed continuous positive airway pressure.
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP — 6 weeks treatment with fixed CPAP
  Other Names: Continuous Positive Airway Pressure
  Arms: Fixed
Device: APAP — 6 weeks of treatment with auto-titrating positive airway pressure
  Other Names: auto-titrating airway pressure
  Arms: auto-titrating

SUMMARY:
The primary objective is to evaluate the relative effectiveness of fixed CPAP in comparison to APAP in reducing arterial blood pressure in patients with resistant hypertension and obstructive sleep apnea (OSA).

The secondary objectives are: a) to evaluate the relative effectiveness of fixed CPAP versus APAP in improving arterial stiffness, sleep-disordered breathing, sleep quality, inflammatory markers and glucose regulation; b) to identify specific characteristic of persons who respond to the two CPAP modalities in order to identify which device is better for each subject.

DETAILED DESCRIPTION:
The confirmatory hypothesis is that subjects with resistant hypertension and OSA will show a greater degree of blood pressure reduction after 6 weeks of treatment with fixed CPAP in comparison to those treated with APAP. Explanatory and exploratory hypotheses are that a greater reduction in arterial stiffness will be noted when compared with the benefit in blood pressure, that reductions in arterial stiffness will be associated with benefits to serum measurements of inflammatory markers and glucose regulation, and that control of sleep apnea and the attendant improvement in sleep quality will be better with fixed CPAP than APAP.

ELIGIBILITY:
Inclusion Criteria:

* Resistant Hypertension
* Moderate Obstructive Sleep Apnea

Exclusion Criteria:

* Creatinine >150 μmol/l
* Systolic blood pressure > 170 mmHg
* Diastolic blood pressure > 105 mmHg
* Secondary cause of hypertension other than OSA
* Treatment within the last 3 months or current treatment for sleep-disordered breathing or some other sleep disorder
* Current treatment or recent treatment within the last 3 months for any other medical condition which has resulted or would be expected to result in a change in blood pressure medications

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2009-12; Primary Completion 2014-01 (Actual); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
24 hour blood pressure. | 6 weeks and 12 weeks after initial intervention

SECONDARY OUTCOMES:
Non-invasive measures of arterial stiffness using applanation tonometry. | 6 weeks and 12 weeks after initial intervention
Standard measures of OSA severity, including AHI and measures of nocturnal oxygenation and sleep quality using polysomnography. | 6 weeks and 12 weeks after initial intervention
Blood tests to assess levels of aldosterone, hsCRP, fasting glucose, HbA1c, and plasma insulin. | 6 weeks and 12 weeks after initial intervention

CONTACTS AND LOCATIONS:
Overall Officials: Stella S Daskalopoulou, MD, MSc, PHd, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; R John Kimoff, MD, FRCP(C), Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (2):
- Canada (2):
  - Royal Victoria Hospital, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec